CLINICAL TRIAL: NCT04856761
Title: A Phase II, Open-Label Study of Capecitabine Versus S-1 as Adjuvant Therapy in Patients With Biliary Tract Carcinoma After Surgical Resection
Brief Title: A Study of Capecitabine Versus S-1 as Adjuvant Therapy in Patients With Biliary Tract Carcinoma After Surgical Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Director, Department of Surgery, Huashan Hospital, Fudan University
Other Study IDs: HUASHAN005
Record Dates: First submitted 2021-04-22; First posted 2021-04-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Biliary Tract Neoplasms; Recurrence; Cholangiocarcinoma; Gall Bladder Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Recurrence; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — S 1 (combination); Tegafur; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor specimen of surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cape Group: In this group, capecitabine was administered at a dose of 1250 mg/m² bid on 14 days of a tri-weekly cycle for 8 cycles.
  Interventions: Drug: Capecitabine
- S-1 Group: In this group, S-1 was administered at a dose of 80-120 mg/day on 14 days of a tri-weekly cycle for 8 cycles.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — S-1 was administered at a dose of 80-120 mg/day on 14 days of a tri-weekly cycle for 8 cycles.
  Other Names: Tegafur
  Groups: S-1 Group
Drug: Capecitabine — Capecitabine was administered at a dose of 1250 mg/m² bid on 14 days of a tri-weekly cycle for 8 cycles.
  Other Names: XELODA
  Groups: Cape Group

SUMMARY:
The purpose of this study is to assess the difference of safety and efficacy about Capecitabine and S-1 for treatment of patients with low-risk of recurrence after BTC surgery.

DETAILED DESCRIPTION:
Patients received curative BTC surgery will be informed about the study. After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be observed for recurrence of BTC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age> 18 years old, and <75 years old.
2. Diagnosis is gallbladder cancer or biliary adenocarcinoma via pathological histology.
3. Patients have received curative surgery of gallbladder cancer or bile duct cancer, and postoperative pathology has confirmed R0 / R1 resection.
4. Ability to comply with the study protocol, in the investigator's judgment.
5. No tumor recurrence before the start of chemotherapy.
6. No fluorouracil drugs were used in the past six months.
7. The main organ function is good, that is, within 14 days before the start of medication, laboratory inspection confirmed that there is sufficient bone marrow function, liver function, renal function, heart function: hemoglobin ≥90g / L; neutral granulocyte count ≥1.5 × 109 / L; platelet ≥ 70 × 109 / L; alt, AST ≤ 3 × ULN (normal value upper limit); total bilirubin ≤ 2.5 × ULN (normal value upper limit)); serum creatinine <1.5 × ULN (normal value upper limit); Serum albumin ≥ 30g / L; coagulation function: PT extended <2s.
8. ECOG score <2.
9. Signed Informed Consent Form.
10. Male and female subjects with potential fertility must agree to adopt high-efficiency contraceptive methods during the study of at least 3 months after receiving the last treatment.

Exclusion Criteria:

1. First chemotherapy start time > 16 postoperatively weeks.
2. Patients with other tumors, or patients with recurrence before chemotherapy;
3. History of allergic with study drugs;
4. History of organ transplantation requires immunosuppressive treatment;
5. Pregnancy or lactation women;
6. Accept the following system treatment within 4 weeks before the start of treatment: cytotoxic treatment, signal conduction inhibitors, immunotherapy, hormone therapy.
7. Participate in other clinical trials within 3 months;
8. Abnormality of the peripheral nervous system (> NCI CTC 1), clinically significant mental abnormalities, have a history of abnormal history of the central nervous system;
9. Electrocardiogram abnormal or clinically obvious heart disease, such as: congestive heart failure, symptomatic coronary heart disease, arrhythmia, clinical manifestations of heart disease, or epasus in the past 12 months; severe infection (> GRADE 2 National Cancer Institute [NCI] -Common Terminology Criteria for AdverSe Events [CTCAE] Version 3.0), sepsis, severe metabolism or diabetes; Digestive ulcer activity period requires treatment, absorption disabilities, diarrhea, intestinal obstruction , Destroyer of the upper deactivated tract integrity;
10. History of HIV infection;
11. Anti-viral treatment cannot be controlled or chronic hepatitis C;
12. Renal failure requires blood or peritoneal dialysis;
13. There are some other serious or unstable diseases or medical, social, sychological states, can endanger the safety of the subject and / or his / her to study the compliance or can prevent patients to participate in clinical research or The assessment of the research results;
14. Refused follow-up in accordance with the requirements set by this research program, as well as refused to sign informed consent.
15. Other factors that may affect patient income and assessment results;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have received curative surgery of pathological diagnosed gallbladder cancer or bile duct cancer.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
RFS, recurrence-free survival | Enrollment to 1 year
  RFS was counted from the enrollment to the date on which disease progression or death was detected, or was censored on the last date when progression-free status was confirmed.

SECONDARY OUTCOMES:
OS, overall survival | Enrollment to 3 years
  OS was calculated from the enrollment to the date of death, or censored on the date of last contact for surviving patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Shanghai, China